CLINICAL TRIAL: NCT04652453
Title: Feasibility, Acceptability, and Barriers to Implementation of a Geriatrics Bundle in the Intensive Care Unit (ACE-ICU)
Brief Title: Feasibility, Acceptability, and Barriers to Implementation of a Geriatrics Bundle in the ICU
Acronym: ACE-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000029410; P30AG021342 (NIH)
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Geriatrics

STUDY DESIGN:
Intervention Model Description: Pre-/Post-Intervention Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-Intervention Group (Geriatrics Bundle) (Experimental): Enrolled participants in the intervention arm will receive all 3 components of the geriatrics bundle: occupational therapy (in addition to physical therapy) upon enrollment in the ICU, a portable amplifying device upon enrollment in the ICU, and a de-prescribing intervention by the ICU pharmacist (in conjunction with the medical team) upon ICU-to-floor transfer.
  Interventions: Other: Geriatrics Bundle
- Pre-Intervention Group (Control) (No Intervention): Participants in the control arm will be enrolled prior to implementation of the geriatrics bundle to gather preliminary data about the secondary outcomes.

INTERVENTIONS:
Other: Geriatrics Bundle — Enrolled participants in the intervention arm will receive all 3 bundle components: occupational therapy (in addition to physical therapy) upon enrollment in the ICU, a portable amplifying device upon enrollment in the ICU, and a de-prescribing intervention by the ICU pharmacist (in conjunction with the medical team) upon ICU-to-floor transfer.
  Arms: Post-Intervention Group (Geriatrics Bundle)

SUMMARY:
Despite the known benefits of geriatric care models among hospitalized older adults outside the intensive care unit (ICU), few studies have addressed the needs of older adults in the ICU; for example, sensory impairment, functional decline, and de-prescribing of potentially inappropriate medications (PIMs) are rarely addressed in routine ICU practice. This pilot study will evaluate the feasibility, acceptability, and barriers to implementation of a geriatrics bundle (occupational therapy, assessment and treatment of hearing impairment, and de-prescribing PIMs) in the ICU.

DETAILED DESCRIPTION:
Outcome 4 was updated 11/8/23.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 65 years
2. Hospitalized in the Medical Intensive Care Unit (MICU) on the York Street campus of Yale-New Haven Hospital.
3. Has not opted out of research

Exclusion Criteria:

1. Unable to provide informed consent and no proxy available
2. Advance directive of "comfort measures only" (CMO) or change to CMO anticipated during this hospital admission
3. Planned discharge to hospice
4. Primary language other than English
5. Tracheostomy with long-term ventilator dependence
6. Patients with non-family conservators (e.g. a lawyer serving as the conservator for the patient)
7. Unable to participate in the OT and hearing impairment interventions due to cognitive status (e.g. advanced dementia, anoxic brain injury, vegetative state, etc) or the need for deep sedation (e.g. if treatment of the critical illness requires deep sedation and neuromuscular blockade, such as in severe ARDS [the acute respiratory distress syndrome])
8. COVID-19 positive
9. Already receiving OT in the ICU

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Ferrante, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 participants and 11 providers
Groups:
- Providers: Providers were surveyed for the acceptability outcome only.
Period: Overall Study
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control) | Providers
Started | 50 | 22 | 11
Completed | 35 | 15 | 11
Not Completed | 15 | 7 | 0
Not completed — Death | 8 | 2 | 0
Not completed — Hospice | 5 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Providers: 11 Providers were surveyed for the acceptability outcome only. Demographics were not collected for the providers.
- Total: Total of all reporting groups
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control) | Providers | Total
Number analyzed (Participants) | 50 | 22 | 11 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Not collected for providers
  years
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 79.48 (7.11) | 76.91 (8.09) |  | 78.69 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    Female | 23 | 12 |  | 35
    Male | 27 | 10 |  | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    White, Non-Hispanic: number analyzed (Participants) | 50 | 22 | 0 | 72
    White, Non-Hispanic | 40 | 18 |  | 58
    White, Hispanic: number analyzed (Participants) | 50 | 22 | 0 | 72
    White, Hispanic | 2 | 0 |  | 2
    Black, non-Hispanic: number analyzed (Participants) | 50 | 22 | 0 | 72
    Black, non-Hispanic | 6 | 3 |  | 9
    Black, Hispanic: number analyzed (Participants) | 50 | 22 | 0 | 72
    Black, Hispanic | 0 | 0 |  | 0
    Hispanic, race not reported: number analyzed (Participants) | 50 | 22 | 0 | 72
    Hispanic, race not reported | 0 | 0 |  | 0
    Non-Hispanic, race not reported: number analyzed (Participants) | 50 | 22 | 0 | 72
    Non-Hispanic, race not reported | 0 | 0 |  | 0
    Asian, non-Hispanic: number analyzed (Participants) | 50 | 22 | 0 | 72
    Asian, non-Hispanic | 2 | 0 |  | 2
    Unknown race and ethnicity: number analyzed (Participants) | 50 | 22 | 0 | 72
    Unknown race and ethnicity | 0 | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 22 | 11 | 83
Highest level of education completed [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    Less than high school: number analyzed (Participants) | 50 | 22 | 0 | 72
    Less than high school | 9 | 3 |  | 12
    High school or equivalent: number analyzed (Participants) | 50 | 22 | 0 | 72
    High school or equivalent | 30 | 8 |  | 38
    2- or 4- year degree: number analyzed (Participants) | 50 | 22 | 0 | 72
    2- or 4- year degree | 6 | 8 |  | 14
    Graduate or post-graduate: number analyzed (Participants) | 50 | 22 | 0 | 72
    Graduate or post-graduate | 4 | 6 |  | 10
Medicaid recipient [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 18 | 6 |  | 24
Marital status [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    Married or living with partner: number analyzed (Participants) | 50 | 22 | 0 | 72
    Married or living with partner | 21 | 13 |  | 34
    Single: number analyzed (Participants) | 50 | 22 | 0 | 72
    Single | 3 | 2 |  | 5
    Divorced or separated: number analyzed (Participants) | 50 | 22 | 0 | 72
    Divorced or separated | 9 | 3 |  | 12
    Widowed: number analyzed (Participants) | 50 | 22 | 0 | 72
    Widowed | 16 | 4 |  | 20
    Other: number analyzed (Participants) | 50 | 22 | 0 | 72
    Other | 1 | 1 |  | 2
Lives alone [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 16 | 4 |  | 20
Respondent [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    Participant: number analyzed (Participants) | 50 | 22 | 0 | 72
    Participant | 34 | 19 |  | 53
    Proxy: number analyzed (Participants) | 50 | 22 | 0 | 72
    Proxy | 16 | 3 |  | 19
Comorbidity count [Median (Inter-Quartile Range); unit: count of comorbidities] — range, 0-10 Population: Not collected for providers
  count of comorbidities
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 3 [2 to 4] | 3.5 [2 to 5] |  | 3 [2 to 4]
Presence of functional disability in any of the 15 activities [Count of Participants; unit: Participants] — The 15 functional activities included seven basic activities of daily living (eating, dressing, bathing, toileting, grooming, getting in and out of a chair, walking around indoors); five instrumental activities of daily living (doing housework, going shopping, preparing a meal, taking medications, managing finances); and three mobility activities (walking a quarter of a mile, climbing stairs, and lifting or carrying heavy objects). A higher score indicates greater disability. Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 37 | 16 |  | 53
Hearing impairment [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 27 | 11 |  | 38
Vision impairment [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 12 | 6 |  | 18
Fall prior to hospitalization [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 22 | 12 |  | 34
Disability in month prior to hospitalization [Median (Inter-Quartile Range); unit: number of activities] — Number of functional activities participant experienced disability (range, 0-15), median (IQR) Population: Not collected for providers
  number of activities
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 4 [1 to 11] | 2.5 [0 to 6] |  | 3 [0 to 8]
Hospitalization in the 6 months prior to admission [Count of Participants; unit: Participants] — Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 33 | 10 |  | 43
History of tobacco use [Count of Participants; unit: Participants] — current or former Population: Not collected for providers
  Participants
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 32 | 15 |  | 47
Clinical Frailty Scale, range 1-7 [Mean (Standard Deviation); unit: score on a scale] — Clinical Frailty Scale (CFS), which measures frailty. The range of scores is 1-7, where a higher score indicates higher frailty (a worse outcome). Population: Not collected for providers
  score on a scale
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 4.87 (1.41) | 4.52 (1.29) |  | 4.76 (1.37)
Muscle strength at baseline, range 0-60 mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Medical Research Council Sum Score (MRC-SS). Strength in each of 6 muscle groups bilaterally is assessed. Each muscle group is scored from 0 (no visible or palpable contraction) to 5 (normal power). If the maneuver was not attempted for a given muscle group, it was assigned a score of zero.The indvidual scores are then summed to make a total score (range, 0-60). Lower scores indicate less strength. There were 13 participants missing the entire MRC-SS assessment in the intervention group and 1 missing in the control group at baseline. Population: Not collected for providers
  units on a scale
    number analyzed (Participants) | 50 | 22 | 0 | 72
    (all) | 46.4 (12.0) | 44.0 (14.2) |  | 45.6 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Bundle Delivery
Description: Feasibility of bundle delivery will be measured by review of electronic medical record (EMR) documentation of each bundle component and a daily-check in with the patient and team. We will determine the proportion of eligible patients receiving each component as well as delivery of the overall bundle. A feasibility threshold of 70% will be used for the individual bundle components, as well as the combined bundle.
Time Frame: From ICU admission to hospital discharge, up to 30 days
Population: Only participants in the geriatric bundle were eligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 50 | 0
Participants | 50 |

2. Primary Outcome: Acceptability of Bundle Delivery
Description: Acceptability of the bundle among providers will be assessed with a survey using a 5-point Likert scale (range 1-5, where 5 indicates that participants strongly agree the bundle is completely acceptable for use in its current form and are comfortable using it).
Time Frame: From ICU admission to hospital discharge, up to 30 days
Population: 11 providers
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Intervention Group (Geriatrics Bundle)
Number analyzed (Participants) | 11
Participants
  Strongly agree | 5
  Agree | 6

3. Primary Outcome: Barriers and Facilitators to Bundle Implementation
Description: Barriers and facilitators to bundle implementation will be assessed using qualitative methods. Separate focus groups were conducted with members of each health care discipline. Focus groups were audio-recorded and transcribed. Content analysis was then used to identify barriers and facilitators to bundle implementation.
Time Frame: From ICU admission to hospital discharge, up to 30 days
Population: Numbers represented here are the number of themes derived from interviews.
Measure: Number; unit: themes
Arm/Group | Post-Intervention Group (Geriatrics Bundle)
Number analyzed (Participants) | 50
themes
  Occupational Therapy Component: Barriers | 7
  Occupational Therapy Component: Facilitators | 3
  Pharmacy Component: Barriers | 5
  Pharmacy Component: Facilitators | 6
  Hearing Amplifier Component: Barriers | 3
  Hearing Amplifier Component: Facilitators | 2

4. Secondary Outcome: Delirium Assessed Using Chart-based Delirium Identification Instrument for ICU (CHART-DEL-ICU)
Description: Incident delirium as measured by the Chart-based Delirium Identification Instrument for ICU (CHART-DEL-ICU). The CHART-DEL-ICU is a validated delirium detection tool for use in critically ill older adults. Charts were manually reviewed and assigned a level of confidence in the detection of delirium for the hospitalization:
  Level of confidence in detection of delirium
  1. Definite (85%+)
  2. Probable (60-85%)
  3. Possible (40-60%)
  4. Uncertain (10-40%)
  5. No evidence (< 10%) Delirium present during the hospitalization = "definite, probable, or possible" Delirium not present during the hospitalization = "uncertain or no evidence" Numbers represented here are participants with delirium.
Time Frame: during hospitalization, up to 128 days
Population: Only patients that proceeded to hospital discharge within 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 41 | 20
Participants | 5 | 7

5. Secondary Outcome: Mobility Level - Highest Level
Description: Data about mobility level during hospitalization will be gathered from the physical therapy and occupational therapy flowsheets. This was scored on a scale of 0-6 with 6 being the highest level of mobility. Presented is the highest score by participants during the hospitalization period.
Time Frame: From ICU admission to hospital discharge, up to 30 days
Population: Only patients that were able to perform these tasks were analyzed, 2 participants in the geriatrics bundle and 1 participant in the control group were not able to be assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 48 | 21
score on a scale | 4.44 (1.13) | 4.38 (1.28)

6. Secondary Outcome: Mobility Level - Level at Discharge
Description: Data about mobility level during hospitalization will be gathered from the physical therapy and occupational therapy flowsheets. This was scored on a scale of 0-6 with 6 being the highest level of mobility. Presented is the participant score at discharge.
Time Frame: From ICU admission to hospital discharge, up to 30 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 48 | 21
score on a scale | 4.10 (1.29) | 4.10 (1.55)

7. Secondary Outcome: Muscle Strength
Description: Manual muscle testing via the 6-point MRC system: Strength in each of 12 muscle groups is assessed via a 6-point system, in which a score of 0=no contraction, 1=flicker of a contraction, 2=active movement with gravity eliminated, 3=active movement against gravity, 4=active movement against gravity and resistance, 5= normal power. The highest possible score is 60, which would indicate maximum muscle strength.
Time Frame: From ICU admission to hospital discharge, up to 30 days
Population: Only participants with data were analyzed; there were 19 participants in the geriatrics bundle group and 5 participants in the control group that were missing these scores at discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 31 | 17
score on a scale | 50.2 (9.0) | 49.6 (14.0)

8. Secondary Outcome: 30-day Functional Outcomes
Description: Participants will be asked whether they were independently able to complete a series of functional activities, including activities of daily living (ADLs), instrumental activities of daily living (IADLs), and mobility activity. Functional activities included seven basic activities of daily living (eating, dressing, bathing, toileting, grooming, getting in and out of a chair, walking around indoors); five instrumental activities of daily living (doing housework, going shopping, preparing a meal, taking medications, managing finances); and three mobility activities (walking a quarter of a mile, climbing stairs, and lifting or carrying heavy objects). A higher count of activities indicates less disability.
Time Frame: 30 days after hospital discharge
Population: Only participants with data were analyzed.
Measure: Median (Inter-Quartile Range); unit: count of activities
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 41 | 21
count of activities | 5 [2 to 12] | 8 [4 to 12]

9. Secondary Outcome: Number of Participants With Hospital Readmissions Within 30 Days
Description: Participants will be asked if they were readmitted to a hospital within 30 days of hospital. The electronic medical record will also be reviewed for readmissions.
Time Frame: 30 days after hospital discharge
Population: Only participants eligible for readmission were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
Number analyzed (Participants) | 35 | 15
Participants | 5 | 3

10. Secondary Outcome: Number of Participants That Reported Use and Perceived Benefit of Amplifying Device After Hospital Discharge
Description: Participants will be asked whether they are still using the portable amplifying device after hospital discharge and whether they perceive benefit from its use. Presented are the qualitative responses summarized as frequencies.
Time Frame: 30 days after hospital discharge
Population: Out of 7 participants that completed the interview. Amplifying device was only provided to the intervention group and not the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Intervention Group (Geriatrics Bundle)
Number analyzed (Participants) | 7
Participants
  Indicate Perceived benefits | 6
  Did Not Indicate Perceived benefits | 1

ADVERSE EVENTS:
Time Frame: up to 30 days after hospital discharge
Description: Adverse events were not tracked for providers as it was not part of the study protocol.
Arm/Group | Post-Intervention Group (Geriatrics Bundle) | Pre-Intervention Group (Control)
All-Cause Mortality (participants affected / at risk) | 8/50 | 2/22
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/22
Other Adverse Events (participants affected / at risk) | 0/50 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT04652453/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04652453/ICF_001.pdf